CLINICAL TRIAL: NCT05025982
Title: Combination of Lymphatico-venular Anastomosis and Liposuction to Treat Cancer-related Lymphedema: Rationale for a Regional Approach
Brief Title: Combination of Lymphatico-venular Anastomosis and Liposuction to Treat Cancer-related Lymphedema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Guido Gabriele, Professor Guido Gabriele, University of Siena
Other Study IDs: combination
Record Dates: First submitted 2021-04-28; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Description of an Effective Surgical Strategy to Treat Cancer-related Lymphedema; Combination of LVA and Liposuction Guarantees Long Lasting Results
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of partecipants: we combined two surgical techniques in the same group of patients
  Interventions: Procedure: combination of lymphaticovenular anastomosis and liposuction

INTERVENTIONS:
Procedure: combination of lymphaticovenular anastomosis and liposuction — Surgeries were carried out under local anesthesia and light sedation.LVA was performed adopting supramicrosurgical technique.Liposuction was performed following completion of the LVA

SUMMARY:
* cooperation of an International team with many years of experience in surgical management of lymphedema
* description of an effective surgical strategy to treat cancer-related lymphedema, a high incidence pathology
* the combination of LVA and liposuction guarantees long lasting results

DETAILED DESCRIPTION:
Cancer-related lymphedema represents one of the major complications of cancer treatment, especially for breast and gynecologic cancers. Moreover, it has high impact on cancer survivors and healthcare systems. Lymphedema management still remains challenging. The better understanding of lymphedema physiopathology as well as the development of sophisticated surgical and diagnostic techniques have led to effective strategies to address lymphedema patients but, despite the considerable interest in international literature, no consensus exist. The combination of LVA and liposuction may represent an effective strategy in treating patients with cancer-related lymphedema, in order to reach a significant decrease in volume and reduction of lymphangitis rate as well as stable results in time. In addition, it has the aim of being minimally invasive and well tolerated by patients

ELIGIBILITY:
Inclusion Criteria: patients affected by secondary lymphedema

* free from cancer disease

Exclusion Criteria:

- persistence of the neoplastic pathology

- patients affected by primary lymphedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with a previous history of cancer who developed secondary lymphedema and are currently free from cancer
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
change in volume | one year
  change in volume of the limb affected by cancer-related lymphedema

CONTACTS AND LOCATIONS:
Locations (1):
- Guido Gabriele, Siena, Italy

IPD SHARING:
Plan to Share IPD: No